CLINICAL TRIAL: NCT03790293
Title: Clinical and Immunological Long-term Follow-up of Patients With Pemphigus Included in the "RITUXIMAB 3" Trial With Medico-economic Evaluation of the Treatment.
Brief Title: Clinical and Immunological Long-term Follow-up of Patients With Pemphigus Included in the "RITUXIMAB 3" Trial
Acronym: LTFURITUX3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/0070/HP
Record Dates: First submitted 2018-10-08; First posted 2018-12-31 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: Patients included and treated in the RITUXIMAB 3 study (NCT00784589):
  * Rituximab in combination with reduced corticosteroids
  * Standard corticosteroid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab (Experimental): Rituximab in combination with reduced corticosteroids is administrated
  Interventions: Drug: Rituximab; Drug: corticosteroids'therapy
- Standard corticosteroid (Active Comparator): Standard corticosteroid is administrated
  Interventions: Drug: corticosteroids'therapy

INTERVENTIONS:
Drug: Rituximab — Patient was enrolled into the RITUXIMAB 3 study in the arm Rituximab in association with low corticosteroids'therapy
  Arms: Rituximab
Drug: corticosteroids'therapy — Patient was enrolled into the RITUXIMAB 3 study in the arm Patient was enrolled into the RITUXIMAB 3 study in the arm standard corticosteroid

SUMMARY:
Pemphigus is an autoimmune disease specific to the skin and mucous membranes characterized by the production of IgG4 isotype autoantibodies (AC) directed mainly against two proteins involved in interkeratinocyte adhesion: desmoglein 1 (Dsg1 ) and desmoglein 3 (Dsg3) (1-3). The binding of auto-AC on these proteins disrupts their adhesion function, resulting in inter-keratinocyte dysjunction called "acantholysis" responsible for the formation of intraepidermal bubbles.

Treatment of pemphigus is typically based on systemic corticosteroids. High doses are usually necessary because of the frequent cortico-resistance of the disease. In recent years, several studies have focused on the treatment of pemphigus with anti-CD20: rituximab. The "Ritux 3" study (NCT00784589), a randomized, multicentre, randomized, non-blind clinical trial involving 90 patients, found that the use of rituximab as first-line therapy in combination with short corticosteroid therapy was extremely effective and that cortisone sparing was thus obtained limited the occurrence of side effects of treatment. On the other hand, this study showed that the 2 rituximab maintenance infusions of 500 mg to M12 and M18 allowed the maintenance of a high rate of complete remission up to the 3rd year of follow-up.

Questions remain to explain the long-term action of rituximab, in particular that of the evolution of these auto-reactive B cells (specific DSG) away from lymphocyte reconstitution B, as well as the evolution of auto-AC. anti-DSG and total IgG CAs, so as to ensure that the disappearance of the auto-reactive compartment is not accompanied by a long-term overall immunosuppression (and therefore a possible risk of infection).

The immunological changes induced in the long term as well as the precise mechanism of action of these treatments and particularly rituximab which allows a complete remission 5 years after treatment in many patients remain little known.

ELIGIBILITY:
Inclusion Criteria:

* Patient included in the RITUXIMAB 3 study
* Major patient who has read and understood the newsletter and signed the consent form

Exclusion Criteria:

* Person deprived of liberty by an administrative or judicial decision
* Person placed under the safeguard of justice
* Person under tutorship or curators
* Pregnant or lactating woman

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-11-17 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Evaluate the occurrence of long-term serious AEs and AEs in patients initially randomized in the rituximab arm and in those who have secondarily received the product during the course of their pemphigus | 1 day: 5 to 7 years after the inclusion into RITUXIMAB 3 study
  Collect of SAE and AE
Evaluate the long-term relapse rate in patients initially randomized in the rituximab arm and in those who have secondarily received the product during the course of their pemphigus | 1 day: 5 to 7 years after the inclusion into RITUXIMAB 3 study
  Collect of relapses

CONTACTS AND LOCATIONS:
Locations (25):
- France (25):
  - Chu Angers, Angers
  - Ap-Hp Avicenne, Bobigny
  - Chu Bordeaux, Bordeaux
  - Chu Brest, Brest
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Ap-Hp Henri Mondor, Créteil
  - Chu Dijon, Dijon
  - Ch Le Mans, Le Mans
  - Chru Lille, Lille
  - Chu Limoges, Limoges
  - Hcl Edouard Herriot, Lyon
  - Hcl Ch Lyon Sud, Lyon
  - Ap-Hm La Timone, Marseille
  - Chu Montpellier, Montpellier
  - Chu Nantes, Nantes
  - Ah-Hp Cochin, Paris
  - Ap-Hp Saint-Louis, Paris
  - Ap-Hp Cochin, Paris
  - Ap-Hp Bichat, Paris
  - Chu Reims, Reims
  - Chu Rennes, Rennes
  - Chu Rouen, Rouen
  - Chu Saint-Etienne, Saint-Etienne
  - Chu Toulouse, Toulouse
  - Chu Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided